CLINICAL TRIAL: NCT05317299
Title: Comparison of the Effects of Different Exercise Types on Lower Extremity Muscle Thickness, Tendon Thickness, Muscle Strength, Proprioception and Balance
Brief Title: Comparison of the Effects of Different Exercise Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilara Özen Oruk (Other)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Sponsor-Investigator, Dilara Özen Oruk, PT, M.Sc., PhD (c) Research Assistant, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 220023/30
Record Dates: First submitted 2022-03-22; First posted 2022-04-07 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: muscle structure; muscle thickness; joint position sense; postural stability

STUDY DESIGN:
Intervention Model Description: Randomized 3 exercise group (RE, PE and HIIT)
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Exercise Group (Active Comparator): During 8 week progressive resistance exercises (three times a week)
  Interventions: Other: 3 different type of exercise
- Plyometric Exercise Group (Active Comparator): During 8 week progressive plyometric exercises (three times a week)
  Interventions: Other: 3 different type of exercise
- High Intensity Interval Training Group (Active Comparator): During 8 week progressive Hight Intensity Interval Training (three times a week)
  Interventions: Other: 3 different type of exercise

INTERVENTIONS:
Other: 3 different type of exercise — Group 1: Resistance Exercise Group 2: Plyometric Exercise Group 3: Hight Intensity Interval Training

SUMMARY:
This study perform to investigate the comparison of the effects of different exercise types on lower extremity muscle thickness, tendon thickness, muscle strength, proprioception and balance.

DETAILED DESCRIPTION:
The choice of exercise type is affected by many different factors. The purpose of exercise and the physical fitness parameter they want to develop gain importance in this choice.

Resistance exercises (RE) specifically designed to increase muscle strength and hypertrophy; Plyometric exercises (PE) based on energy storage of the muscle during the deceleration phase and release of this energy during the acceleration period and high-intensity interval training (HIIT), which is an advanced form of interval training that includes shorter and lighter recovery periods following short to heavy anaerobic exercise are some of the many types of exercises in the literature and practice.

The purpose of the study is investigate the comparison of the effects of different exercise types on lower extremity muscle thickness, tendon thickness, muscle strength, proprioception and balance.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18-30 years old
2. Being a man
3. Volunteering to participate in the study
4. Having a normal BMI (18.5-24.9) according to the World Health Organization criteria

Exclusion Criteria:

1. Having any physical, mental or psychological illness that may affect participation in the study
2. Having a history of trauma to the lower extremity requiring medical, conservative and surgical treatment in the last 6 months
3. Consuming alcohol or pharmaceuticals up to 24 hours before the assessment

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Muscle Thickness assessment with B-mode Ultrasonography | 8 weeks
  Changes of lower extremity muscle thickness
Tendon Thickness assessment with B-mode Ultrasonography | 8 weeks
  Changes of lower extremity tendon thickness
Muscle Strength assessment with manual dinamometer | 8 weeks
  Changes of lower extremity muscle strength
Joint position sense assessment with angle repetition test | 8 weeks
  Changes of lower extremity joint position sense
a kinesthetic ability trainer (Sport KAT Model 650-TS) | 8 weeks
  Changes of static and dynamic balance

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Koçman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided